CLINICAL TRIAL: NCT01860625
Title: A Phase I Clinical, Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of Donepezil Patch in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icure Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IPI-001
Record Dates: First submitted 2013-05-15; First posted 2013-05-23 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- 1(12.5㎠) (Experimental): drug : 9 people, 43.75mg/12.5㎠
  placebo : 3 people, 12.5㎠
  Interventions: Drug: Donepezil patch; Drug: placebo
- 2(25㎠) (Experimental): drug : 9 people, 87.5mg/25㎠
  placebo : 3 people, 25㎠
  Interventions: Drug: Donepezil patch; Drug: placebo
- 3(50㎠) (Experimental): drug : 9 people, 175mg/50㎠
  placebo : 3 people, 50㎠
  Interventions: Drug: Donepezil patch; Drug: placebo

INTERVENTIONS:
Drug: Donepezil patch
Drug: placebo

SUMMARY:
Study of the Safety, tolerability and pharmacokinetics with single dose of donepezil patch in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI : more than 20 ㎏/㎡, less than 26 ㎏/㎡
* Systolic blood pressure : more than 90, less than 140 (mmHg)
* Diastolic blood pressure : more than 60, less than 100 (mmHg)

Exclusion Criteria:

* Evidence of clinically significant, severe, active, or unstable gastrointestinal, renal,hepatic, respiratory, hematological, endocrine, or cardiovascular system disease.
* A history of skin disease or skin graft
* Hypersensitivity to donepezil or piperidine derivatives or any of the excipients.
* A known or suspected history of drug or alcohol dependency or abuse
* Patients who have participated in another clinical study within 60 days.
* Whole blood within 60 days, apheresis within 30 days, transfusion within 30 days
* Heavy caffeine intake(more than 5 units/day)
* Heavy alcohol intake(more than 21 units/week)
* Heavy smoker(more than 10 cigarette/day)
* Abnormal clinical laboratory values which are judged clinically significant by the investigator.
* Any condition that would make the patient or the caregiver, in the opinion of the investigator, unsuitable for the study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
safety and tolerability evaluation | -1d~20d
  evaluation item
  1. adverse event
  2. electrocardiographie
  3. vital sign
  4. physical examination
  5. urine, blood test
  6. skin irritation

SECONDARY OUTCOMES:
pharmacokinetics characteristic evaluation | 1d 0h(before administration), (after administration)4h, 8h, 12h, 24h, 48h, 70h, 72h, 74h, 76h, 80h, 96h, 120h, 144h, 168h, 216h, 264h, 312h
  evaluation item : donepezil conc.
  evaluation variable
  * AUC last, AUC0-∞, Cmax, tmax, t1/2β, CL/F

CONTACTS AND LOCATIONS:
Locations (1):
- ASAN Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi HY, Kim YH, Hong D, Kim SS, Bae KS, Lim HS. Therapeutic dosage assessment based on population pharmacokinetics of a novel single-dose transdermal donepezil patch in healthy volunteers. Eur J Clin Pharmacol. 2015 Aug;71(8):967-77. doi: 10.1007/s00228-015-1875-2. Epub 2015 May 28. PMID 26014587